CLINICAL TRIAL: NCT00651261
Title: A Phase III Randomized, Double-Blind Study of Induction (Daunorubicin/Cytarabine) and Consolidation (High-Dose Cytarabine) Chemotherapy + Midostaurin (PKC412) (IND #101261) or Placebo in Newly Diagnosed Patients < 60 Years of Age With FLT3 Mutated Acute Myeloid Leukemia (AML)
Brief Title: Daunorubicin, Cytarabine, and Midostaurin in Treating Patients With Newly Diagnosed Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CALGB-10603; CALGB-10603; EUDRACT-2006-006852-37; CDR0000590404 (Registry Identifier: Phyisician Data Query)
Record Dates: First submitted 2008-04-01; First posted 2008-04-02 (Estimated); Results first posted 2017-02-06 (Estimated); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Leukemia
Keywords: adult acute basophilic leukemia; adult acute eosinophilic leukemia; adult acute lymphoblastic leukemia; adult acute megakaryoblastic leukemia (M7); adult acute minimally differentiated myeloid leukemia (M0); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myelomonocytic leukemia (M4); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); untreated adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — Cytarabine; Daunorubicin; midostaurin; dexamethasone acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Induction and consolidation chemotherapy plus midostaurin (Experimental): Patients will receive a standard combination of chemotherapy drugs during remission induction therapy that includes cytarabine, daunorubicin, and the experimental drug midostaurin. Depending on the outcome of remission induction treatment, there may be a decision to discontinue the study treatment or a second remission induction cycle may be given. If remission induction therapy is successfully completed, patients will receive four courses of high-dose cytarabine consolidation chemotherapy plus dexamethasone together with the experimental drug midostaurin. All patients will undergo a bone marrow aspiration (and perhaps a biopsy) after the final course of remission consolidation chemotherapy. If the patient continues to respond to the treatment, the patient will receive continuation therapy with midostaurin for twelve (12) months.
  Interventions: Drug: cytarabine; Drug: daunorubicin; Drug: midostaurin; Drug: dexamethasone acetate
- Induction and consolidation chemotherapy plus placebo (Active Comparator): Patients will receive a standard combination of chemotherapy drugs during remission induction therapy that includes cytarabine, daunorubicin, and placebo. Depending on the outcome of remission induction treatment, there may be a decision to discontinue the study treatment or a second remission induction cycle may be given. If remission induction therapy is successfully completed, patients will receive four courses of high-dose cytarabine consolidation chemotherapy plus dexamethasone together with placebo. All patients will undergo a bone marrow aspiration (and perhaps a biopsy) after the final course of remission consolidation chemotherapy. If the patient continues to respond to the treatment, the patient will receive continuation therapy with placebo for twelve (12) months.
  Interventions: Drug: cytarabine; Drug: daunorubicin; Other: placebo; Drug: dexamethasone acetate

INTERVENTIONS:
Drug: cytarabine — Given IV
Drug: daunorubicin — Given IV
Drug: midostaurin — Given orally
  Arms: Induction and consolidation chemotherapy plus midostaurin
Other: placebo — Given orally
  Arms: Induction and consolidation chemotherapy plus placebo
Drug: dexamethasone acetate — ocular medication administration

SUMMARY:
The purpose of this study is to compare the effects, good and/or bad, of a standard chemotherapy regimen for AML that includes the drugs daunorubicin and cytarabine combined with or without midostaurin (also known as PKC412), to find out which is better. This research is being done because it is unknown whether the addition of midostaurin to chemotherapy treatment is better than chemotherapy treatment alone. Midostaurin has been tested in over 400 patients and is being studied in a number of illnesses, including AML, colon cancer, and lung cancer. Midostaurin blocks an enzyme, produced by a gene known as FLT3, that may have a role in the survival and growth of AML cells. Not all leukemia cells will have the abnormal FLT3 gene. This study will focus only on patients with leukemia cells with the abnormal FLT3 gene.

DETAILED DESCRIPTION:
In this study, patients will receive either the experimental agent (midostaurin) or placebo combined with chemotherapy treatment. Patients are stratified according to FLT3 mutation status (internal tandem duplication [ITD] allelic ratio < 0.7 vs ITD allelic ratio ≥ 0.7 vs tandem kinase domain [TKD]). There are three parts to the study treatment: remission induction therapy, remission consolidation therapy and continuation therapy.

Remission Induction Therapy:

* Cytarabine 200 mg/m2/day by continuous intravenous infusion on days 1-7
* Daunorubicin 60 mg/m2/day by intravenous push or short infusion on days 1-3
* Midostaurin 50 mg (two 25 mg capsules) or placebo for midostaurin (2 capsules) twice a day by mouth on days 8-21
* A bone marrow aspiration will be performed in all patients on Day 21 to determine the need for a second induction cycle.

Remission Consolidation (Four Remission Consolidation Cycles):

* High dose cytarabine 3000 mg/m2 will be given by intravenous infusion over 3 hours every 12 hours on days 1, 3 and 5. Serial neurologic evaluation will be performed before and following the infusion of high-dose cytarabine.
* Dexamethasone 0.1% or other corticosteroid ophthalmic solution 2 drops to each eye once daily to begin 6-12 hours prior to the initiation of the cytarabine infusion and to continue for at least 24 hours after the last cytarabine dose.
* Midostaurin 50 mg (two 25 mg capsules) or placebo for midostaurin (2 capsules) twice a day by mouth on days 8-21

Midostaurin/Placebo Continuation Therapy:

* Midostaurin 50 mg (two 25 mg capsules) or placebo for midostaurin (2 capsules) by mouth twice a day for 28 days. Each cycle will be 28 days in length. Continuation therapy with midostaurin/placebo will continue until relapse or for 12 cycles maximum.

The primary and secondary objectives of this study are:

Primary objective:

* To determine if the addition of midostaurin to daunorubicin/cytarabine induction, high-dose cytarabine consolidation, and continuation therapy improves overall survival (OS) in both the mutant FLT3-ITD and FLT3-TKD AML patients

Secondary objectives:

* To compare the overall survival (OS) in the two groups using an analysis in which patients who receive a stem cell transplant are censored at the time of transplant
* To compare the complete response (CR) rate between the two treatment groups
* To compare the event-free survival (EFS) between the two treatment groups
* To compare the disease free survival (DFS) of the two treatment groups
* To compare the disease free survival rate one year after completion of the continuation phase of the two groups
* To assess the toxicity of the experimental combination
* To describe the interaction between treatment outcome and pretreatment characteristics such as age, performance status, white blood cell (WBC) count, morphology, cytogenetics, and molecular and pharmacodynamic features
* To assess the population pharmacokinetics (popPK) of midostaurin and its two major metabolites (CGP52421 and CGP62221). The potential association(s) between PK exposure and FLT3 status, OS, EFS and clinical response will be explored

There is a pharmacokinetic sub-study (CALGB 60706) within CALGB 10603. This embedded companion study must be offered to all patients enrolled on CALGB 10603, although patients may opt not to participate in CALGB 60706.

After study entry, patients are followed periodically for up to 10 years.

ELIGIBILITY:
1. Documentation of Disease:

   * Unequivocal diagnosis of AML ( > 20% blasts in the bone marrow based on the WHO classification), excluding M3 (acute promyelocytic leukemia). Patients with neurologic symptoms suggestive of CNS leukemia are recommended to have a lumbar puncture. Patients whose CSF is positive for AML blasts are not eligible.
   * Documented FLT3 mutation (ITD or point mutation), determined by analysis in a protocol- designated FLT3 screening laboratory.
2. Age Requirement:

   * Age ≥ 18 and < 60 years
3. Prior Therapy:

   * No prior chemotherapy for leukemia or myelodysplasia with the following exceptions:

     * emergency leukapheresis
     * emergency treatment for hyperleukocytosis with hydroxyurea for ≤ 5 days
     * cranial RT for CNS leukostasis (one dose only)
     * growth factor/cytokine support
   * AML patients with a history of antecedent myelodysplasia (MDS) remain eligible for treatment on this trial, but must not have had prior cytotoxic therapy (e.g., azacitidine or decitabine)
   * Patients who have developed therapy related AML after prior RT or chemotherapy for another cancer or disorder are not eligible.
4. Cardiac Function: Patients with symptomatic congestive heart failure are not eligible.
5. Initial Laboratory Value: Total bilirubin < 2.5 x ULN (Upper Limit of Normal)
6. Pregnancy and Nursing Status:

   * Non-pregnant and non-nursing due to the unknown teratogenic potential of midostaurin in humans, pregnant or nursing patients may not be enrolled.
   * Women of childbearing potential must have a negative serum or urine pregnancy test within a sensitivity of at least 50 mIU/mL within 16 days prior to registration.
   * Women of child-bearing potential must either commit to continued abstinence from heterosexual intercourse or commit to TWO acceptable methods of birth control:

     * one highly effective method (eg, IUD, hormonal (non-oral contraceptive), tubal ligation, or partner's vasectomy) and
     * one additional effective method (e.g., latex condom, diaphragm or cervical cap)
   * The two acceptable methods of birth control must be used AT THE SAME TIME, before beginning midostaurin/placebo therapy and continuing for 12 weeks after completion of all therapy.
   * Note that oral contraceptives are not considered a high effective method because of the possibility of a drug interaction with midostaurin.
   * Women of childbearing potential is defined as a sexually active mature woman who has not undergone a hysterectomy or who has not had menses at any time in the preceding 24 consecutive months.
   * Men must agree not to father a child and must use a latex condom during any sexual contact with women of childbearing potential while taking midostaurin/placebo and for 12 weeks after therapy is stopped, even if they have undergone a successful vasectomy.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 717 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard M. Stone, MD, Study Chair — Dana-Farber Cancer Institute
Locations (176):
- United States (170):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California Davis Cancer Center, Sacramento, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Helen and Harry Gray Cancer Center at Hartford Hospital, Hartford, Connecticut
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - H. Lee Moffitt Cancer Center and Research Institute at University of South Florida, Tampa, Florida
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - University of Illinois Cancer Center, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Baystate Regional Cancer Program at D'Amour Center for Cancer Care, Springfield, Massachusetts
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Masonic Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Monter Cancer Center of the North Shore-LIJ Health System, Lake Success, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Tucker Center for Cancer Care at Orange Regional Medical Center, Middletown, New York
  - Winthrop University Hospital, Mineola, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Cleo Craig Cancer Research Clinic, Lawton, Oklahoma
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Penn State Hershey Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Cancer Centers of the Carolinas - Easley, Easley, South Carolina
  - Cancer Centers of the Carolinas - Faris Road, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Grove Commons, Greenville, South Carolina
  - Greenville Hospital Cancer Center, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Self Regional Cancer Center at Self Regional Medical Center, Greenwood, South Carolina
  - Cancer Centers of the Carolinas - Greer Medical Oncology, Greer, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - University of Tennessee Cancer Institute - Memphis, Memphis, Tennessee
  - Tennessee Oncology, PLLC at Sarah Cannon Cancer Center, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Baylor University Medical Center - Houston, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Veterans Affairs Medical Center - Houston, Houston, Texas
  - Mountainview Medical, Berlin Corners, Vermont
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Marshfield Clinic - Chippewa Center, Chippewa Falls, Wisconsin
  - Center for Cancer Treatment & Prevention at Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - D.N. Greenwald Center, Mukwonago, Wisconsin
  - Regional Cancer Center at Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Ministry Saint Clare's Hospital, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
- Canada (6):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Princess Margaret Hospital, Toronto, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - McGill Cancer Centre at McGill University, Montreal, Quebec

REFERENCES:
- [Result] Stone RM, Dohner H, Ehninger G, et al.: CALGB 10603 (RATIFY): A randomized phase III study of induction (daunorubicin/cytarabine) and consolidation (high-dose cytarabine) chemotherapy combined with midostaurin or placebo in treatment-naive patients with FLT3 mutated AML. [Abstract] J Clin Oncol 29 (Suppl 15): A-TPS199, 2011.
- [Derived] Seffernick AE, Mrozek K, Nicolet D, Stone RM, Eisfeld AK, Byrd JC, Archer KJ. High-dimensional genomic feature selection with the ordered stereotype logit model. Brief Bioinform. 2022 Nov 19;23(6):bbac414. doi: 10.1093/bib/bbac414. PMID 36184192
- [Derived] Voso MT, Larson RA, Jones D, Marcucci G, Prior T, Krauter J, Heuser M, Lavorgna S, Nomdedeu J, Geyer SM, Walker A, Wei AH, Sierra J, Sanz MA, Brandwein JM, de Witte TM, Jansen JH, Niederwieser D, Appelbaum FR, Medeiros BC, Tallman MS, Schlenk RF, Ganser A, Amadori S, Cheng Y, Chen Y, Pallaud C, Du L, Piciocchi A, Ehninger G, Byrd J, Thiede C, Dohner K, Stone RM, Dohner H, Bloomfield CD, Lo-Coco F. Midostaurin in patients with acute myeloid leukemia and FLT3-TKD mutations: a subanalysis from the RATIFY trial. Blood Adv. 2020 Oct 13;4(19):4945-4954. doi: 10.1182/bloodadvances.2020002904. PMID 33049054
- [Derived] Walker CJ, Kohlschmidt J, Eisfeld AK, Mrozek K, Liyanarachchi S, Song C, Nicolet D, Blachly JS, Bill M, Papaioannou D, Oakes CC, Giacopelli B, Genutis LK, Maharry SE, Orwick S, Archer KJ, Powell BL, Kolitz JE, Uy GL, Wang ES, Carroll AJ, Stone RM, Byrd JC, de la Chapelle A, Bloomfield CD. Genetic Characterization and Prognostic Relevance of Acquired Uniparental Disomies in Cytogenetically Normal Acute Myeloid Leukemia. Clin Cancer Res. 2019 Nov 1;25(21):6524-6531. doi: 10.1158/1078-0432.CCR-19-0725. Epub 2019 Aug 2. PMID 31375516
- [Derived] Yin J, LaPlant B, Uy GL, Marcucci G, Blum W, Larson RA, Stone RM, Mandrekar SJ. Evaluation of event-free survival as a robust end point in untreated acute myeloid leukemia (Alliance A151614). Blood Adv. 2019 Jun 11;3(11):1714-1721. doi: 10.1182/bloodadvances.2018026112. PMID 31171508
- [Derived] Stein E, Xie J, Duchesneau E, Bhattacharyya S, Vudumula U, Ndife B, Bonifacio G, Guerin A, Li N, Joseph G. Cost Effectiveness of Midostaurin in the Treatment of Newly Diagnosed FLT3-Mutated Acute Myeloid Leukemia in the United States. Pharmacoeconomics. 2019 Feb;37(2):239-253. doi: 10.1007/s40273-018-0732-4. PMID 30382485
- [Derived] Stone RM, Mandrekar SJ, Sanford BL, Laumann K, Geyer S, Bloomfield CD, Thiede C, Prior TW, Dohner K, Marcucci G, Lo-Coco F, Klisovic RB, Wei A, Sierra J, Sanz MA, Brandwein JM, de Witte T, Niederwieser D, Appelbaum FR, Medeiros BC, Tallman MS, Krauter J, Schlenk RF, Ganser A, Serve H, Ehninger G, Amadori S, Larson RA, Dohner H. Midostaurin plus Chemotherapy for Acute Myeloid Leukemia with a FLT3 Mutation. N Engl J Med. 2017 Aug 3;377(5):454-464. doi: 10.1056/NEJMoa1614359. Epub 2017 Jun 23. PMID 28644114
- [Derived] Stone RM, Fischer T, Paquette R, Schiller G, Schiffer CA, Ehninger G, Cortes J, Kantarjian HM, DeAngelo DJ, Huntsman-Labed A, Dutreix C, del Corral A, Giles F. Phase IB study of the FLT3 kinase inhibitor midostaurin with chemotherapy in younger newly diagnosed adult patients with acute myeloid leukemia. Leukemia. 2012 Sep;26(9):2061-8. doi: 10.1038/leu.2012.115. Epub 2012 Apr 27. PMID 22627678

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between May 2008 and October 2001, 3,277 participants were pre-registered. Of those, 900 participants had a documented FLT3 mutation. 717 participants were enrolled onto this study.
Groups:
- Induction and Consolidation Chemotherapy Plus Midostaurin: Patients will receive daunorubicin 60 mg/m^2 by IV push days 1-3 plus cytarabine 200 mg/m^2 IV days 1-7, and midostaurin 50 mg orally twice daily days 8-21. Participants achieving remission will receive four 28 day cycles of high dose cytarabine (3000 mg/m^2) days 1, 3, & 5 and midostaurin at 50 mg orally twice daily days 8-14. Maintenance therapy was given to participants who continued in remission for 12 28-day cycles of midostaurin 50 mg orally twice daily.
- Induction and Consolidation Chemotherapy Plus Placebo: Patients will receive daunorubicin 60 mg/m^2 by IV push days 1-3 plus cytarabine 200 mg/m^2 IV days 1-7, and placebo 50 mg orally twice daily days 8-21. Participants achieving remission will receive four 28 day cycles of high dose cytarabine (3000 mg/m^2) days 1, 3, & 5 and placebo at 50 mg orally twice daily days 8-14. Maintenance therapy was given to participants who continued in remission for 12 28-day cycles of placebo 50 mg orally twice daily.
Period: Overall Study
Arm/Group | Induction and Consolidation Chemotherapy Plus Midostaurin | Induction and Consolidation Chemotherapy Plus Placebo
Started | 360 | 357
Completed | 69 | 51
Not Completed | 291 | 306
Not completed — Adverse Event | 32 | 22
Not completed — Death | 18 | 18
Not completed — Withdrawal by Subject | 22 | 40
Not completed — Induction failure | 24 | 35
Not completed — Disease progression | 58 | 58
Not completed — Alternative therapy | 109 | 107
Not completed — Other disease or participant decisions | 23 | 23
Not completed — Never treated | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Induction and Consolidation Chemotherapy Plus Midostaurin | Induction and Consolidation Chemotherapy Plus Placebo | Total
Number analyzed (Participants) | 360 | 357 | 717
Age, Continuous [Median (Full Range); unit: years] | 47.1 [19 to 59.8] | 48.6 [18 to 60.9] | 47.9 [18.0 to 60.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 186 | 212 | 398
  Male | 174 | 145 | 319
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 7 | 16
  Not Hispanic or Latino | 103 | 107 | 210
  Unknown or Not Reported | 248 | 243 | 491
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 8 | 5 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 9 | 17
  White | 147 | 128 | 275
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 195 | 213 | 408
Region of Enrollment [Number; unit: participants]
  Canada | 4 | 9 | 13
  United States | 117 | 106 | 223
  Germany | 148 | 157 | 305
  Belgium | 3 | 5 | 8
  France | 3 | 2 | 5
  Netherlands | 3 | 2 | 5
  Australia | 0 | 2 | 2
  Spain | 7 | 15 | 22
  Austria | 7 | 5 | 12
  Italy | 61 | 44 | 105
  Czech Republic | 5 | 6 | 11
  Slovakia | 2 | 2 | 4
  Hungary | 0 | 2 | 2
FLT3 mutational subtype [Number; unit: participants] — Mutations in the gene encoding the trans-membrane tyrosine kinase FLT3. FLT3 internal tandem duplications (ITD) mutation which results in a duplication between 3 and greater than 100 amino acids most commonly located in the juxtamembrane region. Tyrosine kinase domain (TKD) point mutations are the remainder of those with FLT3 mutations. FLT3 testing was done centrally.
  participants
    TKD (No ITD) | 81 | 81 | 162
    ITD Allelic ratio <0.7 | 171 | 170 | 341
    ITD Allelic ratio >=0.7 | 108 | 106 | 214

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was defined as the time interval from randomization to death from any cause. The median OS with 95% CI was estimated using the Kaplan-Meier method.
Time Frame: Duration of study (Up to 10 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Induction and Consolidation Chemotherapy Plus Midostaurin | Induction and Consolidation Chemotherapy Plus Placebo
Number analyzed (Participants) | 360 | 357
months | 74.7 [31.5 to NA] — The upper limit was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 25.6 [18.6 to 42.9]
Statistical Analysis 1: Comparison: Induction and Consolidation Chemotherapy Plus Midostaurin vs Induction and Consolidation Chemotherapy Plus Placebo; Test type: Superiority or Other; p = 0.009, 1-sided stratified log-rank; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.63 to 0.96]

2. Secondary Outcome: Event- Free Survival
Description: Event free survival (EFS) was defined as the time from randomization until the earliest qualifying event, including: failure to obtain a CR on or before 60 days of initiation of protocol therapy; relapse; or death from any cause. Patients alive and event free at the time of analysis were censored on the date of last clinical assessment. The median EFS with 95% CI was estimated using the Kaplan-Meier method.
  Due to a higher than expected transplant rate, EFS was promoted to be a key secondary endpoint.
Time Frame: Duration of study (Up to 10 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Induction and Consolidation Chemotherapy Plus Midostaurin | Induction and Consolidation Chemotherapy Plus Placebo
Number analyzed (Participants) | 360 | 357
months | 8.2 [5.4 to 10.7] | 3.0 [1.9 to 5.9]
Statistical Analysis 1: Comparison: Induction and Consolidation Chemotherapy Plus Midostaurin vs Induction and Consolidation Chemotherapy Plus Placebo; Test type: Superiority or Other; p = 0.0024, 1-sided stratified log rank; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.66 to 0.93]

3. Secondary Outcome: Overall Survival, Censoring Participants Who Receive a Stem Cell Transplant at the Time of the Transplant
Description: Overall survival (OS) was defined as the time interval from randomization to death from any cause. Any participants who received a stem cell transplant were censored at the time of transplant. The median OS with 95% CI was estimated using the Kaplan-Meier method.
Time Frame: Duration of study (Up to 10 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Induction and Consolidation Chemotherapy Plus Midostaurin | Induction and Consolidation Chemotherapy Plus Placebo
Number analyzed (Participants) | 360 | 357
months | NA [NA to NA] — The median overall survival with censoring for transplant has not been reached | NA [27.4 to NA] — The median overall survival with censoring for transplant has not been reached

4. Secondary Outcome: Complete Response Rate
Description: Percentage of participants who achieved a complete response (CR). A CR was defined as normalization of blood counts and a marrow showing less than 5% blasts occurring on or before day 60.
Time Frame: Induction therapy (up to 60 days)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction and Consolidation Chemotherapy Plus Midostaurin | Induction and Consolidation Chemotherapy Plus Placebo
Number analyzed (Participants) | 360 | 357
percentage of participants | 59 [54 to 64] | 54 [48 to 59]
Statistical Analysis 1: Comparison: Induction and Consolidation Chemotherapy Plus Midostaurin vs Induction and Consolidation Chemotherapy Plus Placebo; Test type: Superiority or Other; p = 0.15, Fisher Exact

5. Secondary Outcome: Disease-free Survival (DFS)
Description: Disease free survival (DFS) is defined as the time from documentation of first CR at any time to the first of relapse or death from any cause in participants who achieved a CR.
Time Frame: Duration of study (Up to 10 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Induction and Consolidation Chemotherapy Plus Midostaurin | Induction and Consolidation Chemotherapy Plus Placebo
Number analyzed (Participants) | 360 | 357
months | 26.7 [19.4 to NA] — The upper limit was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 15.5 [11.3 to 23.5]
Statistical Analysis 1: Comparison: Induction and Consolidation Chemotherapy Plus Midostaurin vs Induction and Consolidation Chemotherapy Plus Placebo; Test type: Superiority or Other; p = 0.0049, 1-sided stratified log rank

6. Secondary Outcome: DFS Rate One Year After Completing the Planned Continuation Phase
Time Frame: 30 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: 709 participants were evaluated for adverse events.
Arm/Group | Induction and Consolidation Chemotherapy Plus Midostaurin | Induction and Consolidation Chemotherapy Plus Placebo
Serious Adverse Events (participants affected / at risk) | 157/355 | 154/354
Other Adverse Events (participants affected / at risk) | 321/355 | 324/354
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction and Consolidation Chemotherapy Plus Midostaurin (N=355) | Induction and Consolidation Chemotherapy Plus Placebo (N=354)
Blood disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 105 (144) | 110 (152)
Hemoglobin decreased (Blood and lymphatic system disorders) | 154 (237) | 148 (230)
Hemolysis (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphatic disorder (Blood and lymphatic system disorders) | 6 (6) | 4 (4)
Arrhythmia (Cardiac disorders) | 1 (1) | 2 (2)
Asystole (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 6 (6)
Atrial flutter (Cardiac disorders) | 2 (2) | 2 (2)
Atrial tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac disorder (Cardiac disorders) | 4 (4) | 6 (6)
Cardiac pain (Cardiac disorders) | 3 (3) | 1 (1)
Cardiopulmonary arrest (Cardiac disorders) | 0 (0) | 1 (1)
Conduction disorder (Cardiac disorders) | 0 (0) | 2 (2)
Left ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 8 (9) | 7 (7)
Myocardial ischemia (Cardiac disorders) | 3 (3) | 3 (3)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 4 (4) | 5 (5)
Pericarditis (Cardiac disorders) | 3 (3) | 0 (0)
Right ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Sinus arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 17 (20) | 15 (20)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 3 (3)
Ear disorder (Ear and labyrinth disorders) | 1 (1) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 3 (3)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Endocrine disorder (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Conjunctivitis (Eye disorders) | 2 (2) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 1 (1)
Dry eye syndrome (Eye disorders) | 3 (3) | 3 (3)
Eye disorder (Eye disorders) | 8 (9) | 12 (12)
Eye pain (Eye disorders) | 1 (1) | 1 (1)
Eyelid function disorder (Eye disorders) | 0 (0) | 2 (2)
Flashing vision (Eye disorders) | 1 (1) | 2 (2)
Keratitis (Eye disorders) | 5 (6) | 8 (9)
Optic nerve edema (Eye disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 2 (2) | 1 (1)
Retinal detachment (Eye disorders) | 0 (0) | 1 (1)
Scleral disorder (Eye disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 2 (2) | 4 (4)
Watering eyes (Eye disorders) | 2 (2) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 29 (33) | 28 (32)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Anal mucositis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anal pain (Gastrointestinal disorders) | 7 (8) | 5 (5)
Anal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (2) | 2 (2)
Colitis (Gastrointestinal disorders) | 9 (9) | 9 (9)
Colonic hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 16 (18) | 17 (18)
Diarrhea (Gastrointestinal disorders) | 89 (111) | 89 (108)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 1 (1)
Duodenal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 10 (11) | 8 (8)
Dysphagia (Gastrointestinal disorders) | 10 (10) | 10 (12)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 40 (52) | 42 (54)
Endoscopy small intestine abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 2 (2) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Esophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Flatulence (Gastrointestinal disorders) | 7 (8) | 5 (6)
Gastric hemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 10 (12) | 10 (10)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 11 (14) | 7 (7)
Ileal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileal necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (2) | 4 (4)
Intestinal necrosis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Jejunal necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2) | 3 (3)
Mucositis oral (Gastrointestinal disorders) | 23 (23) | 11 (13)
Nausea (Gastrointestinal disorders) | 98 (149) | 91 (126)
Oral hemorrhage (Gastrointestinal disorders) | 5 (6) | 10 (11)
Oral pain (Gastrointestinal disorders) | 5 (5) | 5 (6)
Periodontal disease (Gastrointestinal disorders) | 2 (2) | 1 (1)
Proctitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 3 (3) | 3 (3)
Rectal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 2 (2) | 1 (1)
Salivary gland disorder (Gastrointestinal disorders) | 1 (1) | 2 (2)
Stomach pain (Gastrointestinal disorders) | 8 (12) | 9 (9)
Tooth disorder (Gastrointestinal disorders) | 1 (1) | 2 (2)
Toothache (Gastrointestinal disorders) | 3 (3) | 4 (4)
Typhlitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 70 (101) | 65 (86)
Chest pain (General disorders) | 6 (7) | 11 (12)
Chills (General disorders) | 16 (21) | 16 (24)
Disease progression (General disorders) | 1 (1) | 1 (1)
Edema limbs (General disorders) | 26 (32) | 21 (24)
Facial pain (General disorders) | 2 (2) | 2 (2)
Fatigue (General disorders) | 95 (136) | 98 (130)
Fever (General disorders) | 34 (38) | 33 (38)
Flu-like symptoms (General disorders) | 1 (1) | 1 (1)
General symptom (General disorders) | 11 (14) | 15 (16)
Ill-defined disorder (General disorders) | 1 (1) | 4 (4)
Injection site reaction (General disorders) | 14 (17) | 17 (22)
Localized edema (General disorders) | 5 (5) | 9 (11)
Multi-organ failure (General disorders) | 4 (4) | 5 (5)
Pain (General disorders) | 14 (17) | 18 (24)
Sudden death (General disorders) | 0 (0) | 1 (1)
Visceral edema (General disorders) | 1 (1) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 2 (2)
Hepatobiliary disease (Hepatobiliary disorders) | 4 (4) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 7 (8) | 14 (15)
Immune system disorder (Immune system disorders) | 3 (3) | 3 (4)
Abdominal infection (Infections and infestations) | 1 (1) | 3 (3)
Anal infection (Infections and infestations) | 6 (9) | 5 (5)
Anorectal infection (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bladder infection (Infections and infestations) | 2 (2) | 3 (3)
Bone infection (Infections and infestations) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 3 (4)
Catheter related infection (Infections and infestations) | 29 (39) | 21 (26)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 3 (3) | 2 (2)
Conjunctivitis infective (Infections and infestations) | 4 (4) | 3 (3)
Eye infection (Infections and infestations) | 1 (1) | 1 (1)
Eye infection intraocular (Infections and infestations) | 1 (1) | 0 (0)
Gallbladder infection (Infections and infestations) | 0 (0) | 1 (1)
Gingival infection (Infections and infestations) | 1 (1) | 2 (3)
Hepatic infection (Infections and infestations) | 2 (2) | 3 (3)
Infection (Infections and infestations) | 30 (41) | 26 (33)
Infectious colitis (Infections and infestations) | 8 (8) | 9 (10)
Joint infection (Infections and infestations) | 0 (0) | 2 (2)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Lip infection (Infections and infestations) | 5 (5) | 8 (9)
Lymph gland infection (Infections and infestations) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 1 (1) | 1 (1)
Nail infection (Infections and infestations) | 3 (3) | 0 (0)
Opportunistic infection (Infections and infestations) | 3 (3) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1) | 2 (2)
Otitis media (Infections and infestations) | 0 (0) | 1 (1)
Paranasal sinus infection (Infections and infestations) | 1 (1) | 3 (3)
Penile infection (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 3 (4) | 2 (2)
Phlebitis infective (Infections and infestations) | 2 (2) | 1 (1)
Pleural infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 25 (32) | 35 (39)
Rhinitis infective (Infections and infestations) | 1 (1) | 1 (1)
Salivary gland infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 23 (27) | 16 (17)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 8 (9) | 8 (9)
Small intestine infection (Infections and infestations) | 1 (1) | 0 (0)
Soft tissue infection (Infections and infestations) | 0 (0) | 4 (4)
Splenic infection (Infections and infestations) | 2 (2) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1) | 4 (5)
Upper aerodigestive tract infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 8 (10) | 15 (19)
Vulval infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 4 (4) | 2 (2)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intraoperative complications (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Intraoperative gastrointestinal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intraoperative gastrointestinal injury - Appendix (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intraoperative reproductive tract injury - Ovary (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intraoperative reproductive tract injury - Testis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Kidney anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 9 (15) | 9 (11)
Alanine aminotransferase increased (Investigations) | 35 (41) | 35 (41)
Alkaline phosphatase increased (Investigations) | 8 (8) | 20 (24)
Amylase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 30 (33) | 29 (32)
Blood bilirubin increased (Investigations) | 25 (32) | 36 (42)
CD4 lymphocytes decreased (Investigations) | 1 (3) | 0 (0)
Cardiac troponin T increased (Investigations) | 2 (2) | 1 (1)
Coagulopathy (Investigations) | 8 (14) | 7 (11)
Creatinine increased (Investigations) | 15 (16) | 16 (17)
Electrocardiogram QTc interval prolonged (Investigations) | 17 (22) | 19 (22)
Fibrinogen decreased (Investigations) | 2 (2) | 7 (7)
Gamma-glutamyltransferase increased (Investigations) | 19 (25) | 22 (32)
INR increased (Investigations) | 8 (10) | 5 (5)
Laboratory test abnormal (Investigations) | 18 (33) | 28 (47)
Leukocyte count decreased (Investigations) | 41 (66) | 47 (78)
Lipase increased (Investigations) | 2 (2) | 1 (1)
Lymphocyte count decreased (Investigations) | 22 (30) | 36 (56)
Neutrophil count decreased (Investigations) | 145 (227) | 146 (224)
Platelet count decreased (Investigations) | 155 (239) | 146 (227)
Serum cholesterol increased (Investigations) | 1 (1) | 0 (0)
Weight gain (Investigations) | 3 (3) | 3 (3)
Weight loss (Investigations) | 1 (1) | 11 (13)
Acidosis (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 21 (30) | 26 (29)
Blood glucose increased (Metabolism and nutrition disorders) | 17 (23) | 22 (31)
Blood uric acid increased (Metabolism and nutrition disorders) | 6 (10) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Serum albumin decreased (Metabolism and nutrition disorders) | 19 (28) | 22 (26)
Serum calcium decreased (Metabolism and nutrition disorders) | 20 (25) | 26 (30)
Serum calcium increased (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Serum glucose decreased (Metabolism and nutrition disorders) | 1 (1) | 2 (3)
Serum magnesium decreased (Metabolism and nutrition disorders) | 15 (19) | 15 (22)
Serum phosphate decreased (Metabolism and nutrition disorders) | 7 (9) | 12 (13)
Serum potassium decreased (Metabolism and nutrition disorders) | 31 (37) | 47 (53)
Serum potassium increased (Metabolism and nutrition disorders) | 8 (9) | 4 (4)
Serum sodium decreased (Metabolism and nutrition disorders) | 20 (22) | 20 (22)
Serum sodium increased (Metabolism and nutrition disorders) | 5 (5) | 5 (5)
Serum triglycerides increased (Metabolism and nutrition disorders) | 3 (4) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 6 (6)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 15 (19) | 13 (13)
Bone pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 4 (5)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 4 (5)
Neck pain (Musculoskeletal and connective tissue disorders) | 7 (8) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6) | 6 (9)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 3 (3)
Depressed level of consciousness (Nervous system disorders) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 19 (23) | 20 (25)
Dysgeusia (Nervous system disorders) | 4 (4) | 7 (9)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 41 (54) | 42 (63)
Intracranial hemorrhage (Nervous system disorders) | 3 (3) | 6 (6)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 2 (2) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Neurological disorder NOS (Nervous system disorders) | 9 (11) | 4 (4)
Nystagmus (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (5) | 6 (11)
Seizure (Nervous system disorders) | 1 (1) | 1 (1)
Speech disorder (Nervous system disorders) | 4 (4) | 1 (1)
Syncope (Nervous system disorders) | 6 (6) | 4 (4)
Syncope vasovagal (Nervous system disorders) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 4 (4) | 3 (3)
Agitation (Psychiatric disorders) | 3 (5) | 3 (3)
Anxiety (Psychiatric disorders) | 5 (5) | 9 (11)
Confusion (Psychiatric disorders) | 4 (4) | 3 (3)
Depression (Psychiatric disorders) | 2 (2) | 12 (12)
Euphoria (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 11 (14) | 7 (11)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1)
Psychosis (Psychiatric disorders) | 4 (4) | 2 (2)
Bladder hemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Cystitis (Renal and urinary disorders) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Renal and urinary disorders) | 2 (2) | 1 (1)
Hemorrhage urinary tract (Renal and urinary disorders) | 2 (2) | 6 (6)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 13 (13) | 9 (9)
Renal hemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral pain (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2) | 3 (3)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 15 (21) | 11 (15)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Penile pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Perineal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Reproductive tract disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine hemorrhage (Reproductive system and breast disorders) | 4 (5) | 3 (4)
Vaginal hemorrhage (Reproductive system and breast disorders) | 5 (5) | 9 (9)
Vaginal mucositis (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Vaginal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 5 (5)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (21) | 19 (20)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 20 (22) | 24 (24)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 24 (26) | 22 (24)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 12 (12)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngoscopy abnormal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 11 (12)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 8 (8)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 27 (28) | 17 (19)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 12 (12) | 9 (9)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Retinoic acid syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (8) | 4 (4)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (8) | 7 (7)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 2 (4) | 5 (5)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 35 (45) | 34 (52)
Pruritus (Skin and subcutaneous tissue disorders) | 11 (13) | 12 (13)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 59 (70) | 66 (71)
Skin disorder (Skin and subcutaneous tissue disorders) | 23 (28) | 23 (30)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Sweating (Skin and subcutaneous tissue disorders) | 14 (19) | 14 (15)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (4)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 14 (17) | 13 (17)
Hemorrhage (Vascular disorders) | 14 (19) | 12 (13)
Hot flashes (Vascular disorders) | 1 (1) | 2 (2)
Hypertension (Vascular disorders) | 13 (13) | 11 (11)
Hypotension (Vascular disorders) | 25 (26) | 19 (22)
Lymphangitic streak (Vascular disorders) | 0 (0) | 1 (1)
Lymphedema (Vascular disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 6 (7) | 7 (7)
Thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Vascular disorder (Vascular disorders) | 2 (2) | 2 (2)
Vasculitis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction and Consolidation Chemotherapy Plus Midostaurin (N=355) | Induction and Consolidation Chemotherapy Plus Placebo (N=354)
Blood disorder (Blood and lymphatic system disorders) | 5 (11) | 4 (6)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 246 (422) | 238 (394)
Hemoglobin decreased (Blood and lymphatic system disorders) | 312 (1059) | 311 (940)
Lymph node pain (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Lymphatic disorder (Blood and lymphatic system disorders) | 10 (13) | 9 (11)
Arrhythmia (Cardiac disorders) | 1 (1) | 4 (4)
Atrial fibrillation (Cardiac disorders) | 3 (3) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1)
Atrial tachycardia (Cardiac disorders) | 1 (3) | 1 (1)
Cardiac disorder (Cardiac disorders) | 8 (12) | 13 (17)
Cardiac pain (Cardiac disorders) | 4 (6) | 1 (1)
Cardiac valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Conduction disorder (Cardiac disorders) | 1 (1) | 2 (2)
Left ventricular failure (Cardiac disorders) | 6 (6) | 5 (9)
Myocardial ischemia (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 3 (3) | 5 (13)
Pericardial effusion (Cardiac disorders) | 7 (8) | 1 (1)
Pericarditis (Cardiac disorders) | 2 (2) | 1 (1)
Premature ventricular contractions (Cardiac disorders) | 1 (3) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 10 (10) | 5 (15)
Sinus tachycardia (Cardiac disorders) | 11 (13) | 23 (29)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 2 (7)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Ventricular arrhythmia (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular bigeminy (Cardiac disorders) | 1 (2) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Ear disorder (Ear and labyrinth disorders) | 5 (5) | 3 (3)
Ear pain (Ear and labyrinth disorders) | 5 (6) | 6 (6)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 2 (2)
External ear pain (Ear and labyrinth disorders) | 3 (3) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 2 (4) | 2 (2)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 3 (3) | 2 (2)
Endocrine disorder (Endocrine disorders) | 1 (1) | 2 (2)
Hyperthyroidism (Endocrine disorders) | 2 (7) | 1 (3)
Hypothyroidism (Endocrine disorders) | 2 (2) | 2 (5)
Cataract (Eye disorders) | 1 (9) | 0 (0)
Conjunctivitis (Eye disorders) | 7 (7) | 4 (5)
Dry eye syndrome (Eye disorders) | 5 (7) | 10 (12)
Eye disorder (Eye disorders) | 21 (28) | 16 (19)
Eye pain (Eye disorders) | 5 (5) | 5 (5)
Eyelid function disorder (Eye disorders) | 0 (0) | 1 (1)
Flashing vision (Eye disorders) | 1 (1) | 4 (5)
Keratitis (Eye disorders) | 14 (17) | 9 (14)
Optic nerve disorder (Eye disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 2 (3) | 4 (4)
Vision blurred (Eye disorders) | 5 (8) | 4 (7)
Vitreous hemorrhage (Eye disorders) | 1 (1) | 2 (2)
Watering eyes (Eye disorders) | 4 (7) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 6 (15) | 10 (11)
Abdominal pain (Gastrointestinal disorders) | 57 (78) | 67 (84)
Anal exam abnormal (Gastrointestinal disorders) | 0 (0) | 3 (3)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 2 (2) | 3 (3)
Anal mucositis (Gastrointestinal disorders) | 2 (2) | 2 (3)
Anal pain (Gastrointestinal disorders) | 12 (15) | 6 (8)
Anal ulcer (Gastrointestinal disorders) | 1 (1) | 3 (3)
Ascites (Gastrointestinal disorders) | 1 (1) | 1 (1)
Colitis (Gastrointestinal disorders) | 7 (9) | 12 (18)
Colonic hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 50 (86) | 60 (83)
Dental prosthesis user (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 228 (432) | 219 (310)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 22 (36) | 16 (17)
Dysphagia (Gastrointestinal disorders) | 6 (6) | 10 (10)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 112 (178) | 112 (169)
Endoscopy large bowel abnormal (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Esophageal mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 1 (1) | 3 (3)
Esophageal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 3 (3) | 4 (4)
Flatulence (Gastrointestinal disorders) | 10 (20) | 7 (8)
Gastric hemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastric mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 3 (3) | 4 (4)
Gastrointestinal disorder (Gastrointestinal disorders) | 28 (35) | 26 (29)
Gastrointestinal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroscopy abnormal (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gingival pain (Gastrointestinal disorders) | 3 (3) | 4 (4)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (3)
Hemorrhoids (Gastrointestinal disorders) | 28 (36) | 21 (25)
Ileal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 2 (3) | 3 (3)
Large intestinal mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 49 (59) | 31 (36)
Nausea (Gastrointestinal disorders) | 258 (807) | 226 (449)
Oesophagoscopy abnormal (Gastrointestinal disorders) | 2 (2) | 1 (1)
Oral hemorrhage (Gastrointestinal disorders) | 12 (13) | 18 (27)
Oral pain (Gastrointestinal disorders) | 8 (10) | 11 (11)
Periodontal disease (Gastrointestinal disorders) | 4 (6) | 7 (7)
Peritoneal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctoscopy abnormal (Gastrointestinal disorders) | 3 (3) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 7 (8) | 5 (7)
Rectal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 5 (6) | 2 (2)
Salivary gland disorder (Gastrointestinal disorders) | 0 (0) | 2 (2)
Small intestinal mucositis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Stomach pain (Gastrointestinal disorders) | 34 (43) | 27 (32)
Tooth development disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 6 (6) | 2 (2)
Toothache (Gastrointestinal disorders) | 9 (11) | 10 (10)
Typhlitis (Gastrointestinal disorders) | 3 (3) | 4 (4)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 188 (376) | 168 (259)
Chest pain (General disorders) | 15 (17) | 20 (28)
Chills (General disorders) | 22 (26) | 17 (21)
Disease progression (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 33 (43) | 39 (56)
Facial pain (General disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 221 (522) | 220 (474)
Fever (General disorders) | 72 (110) | 69 (107)
Flu-like symptoms (General disorders) | 5 (5) | 2 (2)
Gait abnormal (General disorders) | 1 (1) | 0 (0)
General symptom (General disorders) | 15 (18) | 17 (25)
Hypothermia (General disorders) | 1 (1) | 0 (0)
Ill-defined disorder (General disorders) | 3 (4) | 4 (4)
Injection site reaction (General disorders) | 20 (25) | 23 (34)
Localized edema (General disorders) | 16 (16) | 14 (19)
Pain (General disorders) | 40 (55) | 33 (44)
Visceral edema (General disorders) | 2 (2) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Gallbladder pain (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatobiliary disease (Hepatobiliary disorders) | 4 (16) | 4 (5)
Cytokine release syndrome (Immune system disorders) | 1 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 36 (41) | 30 (41)
Immune system disorder (Immune system disorders) | 12 (14) | 9 (14)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Anal infection (Infections and infestations) | 8 (9) | 8 (12)
Anorectal infection (Infections and infestations) | 2 (3) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2)
Bladder infection (Infections and infestations) | 8 (13) | 10 (11)
Bone infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 7 (9) | 6 (6)
Catheter related infection (Infections and infestations) | 55 (74) | 43 (54)
Cecal infection (Infections and infestations) | 1 (1) | 1 (2)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 4 (4) | 4 (4)
Conjunctivitis infective (Infections and infestations) | 8 (10) | 5 (7)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 2 (2) | 0 (0)
Gastric infection (Infections and infestations) | 1 (1) | 2 (3)
Gingival infection (Infections and infestations) | 5 (6) | 3 (3)
Hepatic infection (Infections and infestations) | 3 (3) | 5 (14)
Infection (Infections and infestations) | 57 (100) | 60 (99)
Infectious colitis (Infections and infestations) | 5 (7) | 5 (5)
Kidney infection (Infections and infestations) | 2 (2) | 1 (1)
Lip infection (Infections and infestations) | 17 (22) | 21 (29)
Lymph gland infection (Infections and infestations) | 1 (1) | 3 (4)
Mediastinal infection (Infections and infestations) | 1 (1) | 0 (0)
Mucosal infection (Infections and infestations) | 2 (2) | 0 (0)
Nail infection (Infections and infestations) | 3 (4) | 2 (2)
Opportunistic infection (Infections and infestations) | 4 (5) | 9 (14)
Otitis media (Infections and infestations) | 2 (3) | 0 (0)
Paranasal sinus infection (Infections and infestations) | 2 (2) | 1 (1)
Penile infection (Infections and infestations) | 2 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 5 (5) | 7 (7)
Phlebitis infective (Infections and infestations) | 3 (5) | 2 (2)
Pneumonia (Infections and infestations) | 36 (53) | 36 (45)
Rhinitis infective (Infections and infestations) | 6 (12) | 6 (7)
Scrotal infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 26 (29) | 20 (23)
Sinusitis (Infections and infestations) | 7 (7) | 5 (6)
Skin infection (Infections and infestations) | 22 (24) | 15 (19)
Soft tissue infection (Infections and infestations) | 2 (2) | 1 (1)
Splenic infection (Infections and infestations) | 1 (1) | 2 (9)
Tooth infection (Infections and infestations) | 4 (4) | 4 (5)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Upper aerodigestive tract infection (Infections and infestations) | 0 (0) | 4 (4)
Upper respiratory infection (Infections and infestations) | 11 (17) | 8 (14)
Ureteritis (Infections and infestations) | 4 (6) | 4 (6)
Urinary tract infection (Infections and infestations) | 15 (17) | 15 (19)
Vaginal infection (Infections and infestations) | 5 (6) | 8 (12)
Viral hepatitis (Infections and infestations) | 1 (1) | 0 (0)
Vulval infection (Infections and infestations) | 2 (2) | 0 (0)
Vulvitis (Infections and infestations) | 0 (0) | 2 (2)
Wound infection (Infections and infestations) | 3 (3) | 3 (3)
Bruising (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Device complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Injury to inferior vena cava (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury to jugular vein (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intraoperative complications (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intraoperative gastrointestinal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intraoperative gastrointestinal injury - Teeth (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intraoperative head and neck injury - Neck NOS (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intraoperative ocular injury - Lens (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Tracheostomy site bleeding (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vaginal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 9 (15) | 6 (6)
Venous injury - Extremity-lower (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 26 (36) | 22 (27)
Alanine aminotransferase increased (Investigations) | 88 (312) | 83 (184)
Alkaline phosphatase increased (Investigations) | 30 (60) | 29 (55)
Amylase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 60 (201) | 56 (102)
Blood bilirubin increased (Investigations) | 49 (86) | 60 (104)
Cardiac troponin T increased (Investigations) | 1 (1) | 1 (1)
Coagulopathy (Investigations) | 7 (8) | 10 (14)
Creatinine increased (Investigations) | 13 (18) | 15 (25)
Electrocardiogram QTc interval prolonged (Investigations) | 45 (81) | 36 (48)
Fibrinogen decreased (Investigations) | 12 (14) | 8 (10)
Forced expiratory volume decreased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 25 (55) | 34 (57)
INR increased (Investigations) | 9 (11) | 12 (12)
Laboratory test abnormal (Investigations) | 31 (53) | 41 (81)
Leukocyte count decreased (Investigations) | 79 (240) | 92 (204)
Lymphocyte count decreased (Investigations) | 69 (195) | 71 (158)
Neutrophil count decreased (Investigations) | 308 (952) | 308 (879)
Platelet count decreased (Investigations) | 311 (1131) | 313 (1020)
Serum cholesterol increased (Investigations) | 0 (0) | 5 (10)
Weight gain (Investigations) | 15 (26) | 6 (11)
Weight loss (Investigations) | 9 (12) | 10 (12)
Alkalosis (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 30 (40) | 40 (50)
Blood glucose increased (Metabolism and nutrition disorders) | 72 (202) | 59 (134)
Blood uric acid increased (Metabolism and nutrition disorders) | 21 (42) | 15 (23)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 2 (5)
Iron overload (Metabolism and nutrition disorders) | 0 (0) | 2 (4)
Serum albumin decreased (Metabolism and nutrition disorders) | 56 (101) | 56 (80)
Serum calcium decreased (Metabolism and nutrition disorders) | 58 (88) | 56 (79)
Serum calcium increased (Metabolism and nutrition disorders) | 6 (11) | 1 (2)
Serum glucose decreased (Metabolism and nutrition disorders) | 6 (8) | 9 (10)
Serum magnesium decreased (Metabolism and nutrition disorders) | 30 (48) | 32 (65)
Serum magnesium increased (Metabolism and nutrition disorders) | 7 (8) | 3 (3)
Serum phosphate decreased (Metabolism and nutrition disorders) | 27 (31) | 27 (40)
Serum potassium decreased (Metabolism and nutrition disorders) | 79 (117) | 74 (112)
Serum potassium increased (Metabolism and nutrition disorders) | 5 (5) | 5 (6)
Serum sodium decreased (Metabolism and nutrition disorders) | 48 (63) | 51 (64)
Serum sodium increased (Metabolism and nutrition disorders) | 8 (8) | 8 (9)
Serum triglycerides increased (Metabolism and nutrition disorders) | 1 (1) | 4 (5)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 2 (2) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 (67) | 16 (25)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 46 (74) | 34 (53)
Bone pain (Musculoskeletal and connective tissue disorders) | 19 (32) | 21 (37)
Buttock pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 6 (9) | 3 (4)
Joint disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint range of motion decreased lumbar spine (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 6 (6) | 4 (4)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 13 (19) | 6 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 13 (24) | 16 (19)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 16 (18) | 9 (9)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 30 (39) | 17 (23)
Upper extremity dysfunction (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myelodysplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (2)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 2 (2) | 10 (11)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 2 (2) | 3 (3)
Dizziness (Nervous system disorders) | 44 (64) | 43 (55)
Dysgeusia (Nervous system disorders) | 5 (5) | 11 (14)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (5)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 2 (5)
Headache (Nervous system disorders) | 105 (218) | 85 (143)
Intracranial hemorrhage (Nervous system disorders) | 1 (1) | 2 (2)
Memory impairment (Nervous system disorders) | 2 (4) | 1 (2)
Neuralgia (Nervous system disorders) | 2 (2) | 3 (6)
Neurological disorder NOS (Nervous system disorders) | 17 (22) | 7 (7)
Olfactory nerve disorder (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 2 (12) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 6 (21) | 11 (26)
Pyramidal tract syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Speech disorder (Nervous system disorders) | 1 (16) | 1 (1)
Syncope (Nervous system disorders) | 8 (9) | 6 (6)
Syncope vasovagal (Nervous system disorders) | 2 (3) | 7 (9)
Tremor (Nervous system disorders) | 5 (8) | 4 (4)
Agitation (Psychiatric disorders) | 4 (4) | 3 (3)
Anxiety (Psychiatric disorders) | 16 (21) | 18 (32)
Confusion (Psychiatric disorders) | 4 (5) | 4 (4)
Depression (Psychiatric disorders) | 14 (26) | 24 (50)
Euphoria (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 30 (47) | 20 (35)
Personality change (Psychiatric disorders) | 0 (0) | 1 (1)
Psychosis (Psychiatric disorders) | 1 (1) | 1 (1)
Bladder hemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Bladder pain (Renal and urinary disorders) | 3 (5) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 2 (2) | 0 (0)
Cystitis (Renal and urinary disorders) | 5 (6) | 7 (8)
Hemoglobin urine positive (Renal and urinary disorders) | 0 (0) | 1 (1)
Hemorrhage urinary tract (Renal and urinary disorders) | 2 (2) | 4 (4)
Kidney pain (Renal and urinary disorders) | 1 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (3) | 1 (1)
Renal failure (Renal and urinary disorders) | 3 (3) | 1 (1)
Urethral obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral pain (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 4 (9)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1) | 2 (3)
Urine discoloration (Renal and urinary disorders) | 0 (0) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 11 (12) | 10 (11)
Breast pain (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Gynecomastia (Reproductive system and breast disorders) | 1 (1) | 1 (3)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Perineal pain (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Reproductive tract disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine hemorrhage (Reproductive system and breast disorders) | 8 (12) | 6 (7)
Uterine pain (Reproductive system and breast disorders) | 1 (1) | 3 (3)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 1 (2)
Vaginal hemorrhage (Reproductive system and breast disorders) | 16 (17) | 17 (24)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Vaginal mucositis (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Vaginal pain (Reproductive system and breast disorders) | 1 (1) | 2 (2)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 8 (14)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 38 (57) | 41 (51)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 28 (33) | 29 (30)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 55 (63) | 46 (62)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 11 (11)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3)
Laryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Laryngoscopy abnormal (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (6)
Pharyngeal examination abnormal (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 28 (35) | 25 (30)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 6 (6)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 23 (33) | 33 (40)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 17 (23) | 21 (31)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (10) | 6 (9)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 11 (13) | 9 (12)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 8 (9) | 9 (11)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 67 (89) | 51 (68)
Photosensitivity (Skin and subcutaneous tissue disorders) | 3 (5) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 25 (31) | 31 (41)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 201 (358) | 200 (317)
Skin disorder (Skin and subcutaneous tissue disorders) | 44 (67) | 42 (58)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (3) | 3 (4)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Skin striae (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 5 (6) | 6 (8)
Sweating (Skin and subcutaneous tissue disorders) | 30 (50) | 19 (32)
Urticaria (Skin and subcutaneous tissue disorders) | 6 (7) | 5 (5)
Flushing (Vascular disorders) | 0 (0) | 2 (3)
Hematoma (Vascular disorders) | 32 (40) | 34 (39)
Hemorrhage (Vascular disorders) | 15 (22) | 31 (33)
Hot flashes (Vascular disorders) | 2 (4) | 4 (4)
Hypertension (Vascular disorders) | 15 (21) | 13 (25)
Hypotension (Vascular disorders) | 32 (37) | 32 (36)
Lymphedema (Vascular disorders) | 0 (0) | 1 (1)
Lymphocele (Vascular disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 13 (19) | 15 (17)
Thrombosis (Vascular disorders) | 6 (6) | 3 (3)
Vascular disorder (Vascular disorders) | 0 (0) | 4 (4)
Vasculitis (Vascular disorders) | 2 (2) | 0 (0)
Visceral arterial ischemia (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less